CLINICAL TRIAL: NCT07228507
Title: Video-based Educational Intervention on Healthcare Professionals' Knowledge of Relative Energy Deficiency in Sport
Brief Title: Video Intervention of Relative Energy Deficiency in Sport
Acronym: Video_REDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Susana Gil, Principal Investigator, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: M10_2024_104
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Female Athlete Triad; Relative Energy Deficiency in Sport; Knowledge
Keywords: Knowledge; Female Athlete Triad; Relative Energy Deficiency in sport
MeSH Terms: conditions — Female Athlete Triad Syndrome; Relative Energy Deficiency in Sport

STUDY DESIGN:
Masking Description: Participants were randomized (in a 1:1 ratio) by an online tool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational video (Experimental): Participants attend an educational video and complete the questionnaire pre- and post-intervention.
  Interventions: Other: Behavioral: Educational Program on Female Athlete Triad and Relative Energy Deficiency in Sport (RED-S)
- Control (No Intervention): Participants complete the same questionnaire at baseline and follow-up without receiving the educational video

INTERVENTIONS:
Other: Behavioral: Educational Program on Female Athlete Triad and Relative Energy Deficiency in Sport (RED-S) — Participants in the intervention arm attended an educational session designed to improve knowledge about the Female Athlete Triad and REDs, focusing on definition, low energy availability, menstrual function, and bone health.
  Arms: Educational video

SUMMARY:
The Female and Male Athlete Triad (Triad) and Relative Energy Deficiency in Sport (REDs) are multifactorial conditions often under-recognized by healthcare professionals. Improving provider awareness is essential for early detection and multidisciplinary management in sport medicine. Thus, the objective was to assess the effectiveness of a brief online educational video in improving knowledge, attitudes, and perceived confidence toward the Triad and REDs among Spanish healthcare professionals.

DETAILED DESCRIPTION:
The objective was to assess the effectiveness of a brief online educational video in improving knowledge, attitudes, and perceived confidence toward the Triad and REDs among Spanish healthcare professionals.

Design: Randomized controlled educational trial. A total of 200 Spanish healthcare professionals (physicians, nurses, and physiotherapists) were randomized 1:1 into an intervention group (VG) and a control group (CG). The VG received access to an 18-minute YouTube-based educational video titled "Triad of the Female Athlete and RED-S". The CG did not have access to the video until the study was completed. Both completed a validated 16-question questionnaire before and after the intervention.

The Primary Outcome Measure was the change in knowledge score about the Female/Male Athlete Triad and REDs. Secondary outcomes included questions from the definition group (questions 1 and 3), low energy availability group (questions 2, 4, 5, 10, 14, 15 and 16), the menstrual health group (questions 6,9,11 and 13) and the bone health group (questions 7,8 and 12)

Descriptive analyses were conducted to determine means, standard deviations, frequencies, and percentages. A two-way repeated-measures ANOVA was performed after verifying the statistical assumptions required for this methodology. Outliers were examined using the first and third quartiles and the interquartile range. Participants with a total score ≤4 were excluded from the analysis to preserve the reliability and validity of the data and to ensure that statistical analyses reflected only responses with adequate informational content consistent with the study conditions. Data normality was assessed through Q-Q plots and the Shapiro-Wilk test. The effects of the group factor (VG vs. CG), the time factor (pre- vs. post-test), and their interaction were analysed, considering a 95% confidence interval (p ≤ 0.05).

Knowledge Questions

1. What do you consider to be the three components of the Female Athlete Triad?
2. Low energy availability in a person occurs when the energy to maintain the functions required by the human body to preserve health and optimal performance is insufficient.
3. What is the main factor that would cause REDs?
4. Low energy availability could be associated with a decrease in carbohydrate intake.
5. There may be low energy availability without changes in weight or body mass index.
6. Menarche in adolescents after the age of 15 is normal if they engage in intense physical activity.
7. At what age does peak bone mineral density occur in women?
8. Osteopenia in adolescent girls or young adult women can be reversed if, in adulthood, they reduce the intensity or volume of their physical activity.
9. In a physically active woman, secondary amenorrhea can be considered normal if she engages in intense sport.
10. Menstrual disorders in physically active women are a risk factor for having low bone mineral density.
11. Low energy availability can cause secondary amenorrhea in physically active women.
12. In physically active women, menstrual cycle alterations or amenorrhea are indicators of intense training.
13. In physically active women, stress fractures may occur at a higher rate in women with prolonged amenorrhea than in eumenorrheic women.
14. Low energy availability can affect an athlete's recovery.
15. Low energy availability can increase performance (strength, speed, power).
16. After performing intense exercise, the basis of caloric intake should be...

ELIGIBILITY:
Inclusion Criteria:

* Registered in a health professional association in Spain (medicine, nursing, or physiotherapy).
* Voluntary participation and completion of the baseline questionnaire.
* Consent to provide an email address for communication and randomization

Exclusion Criteria:

* Not to be registered in a health professional association in Spain (medicine, nursing, or physiotherapy).
* Incomplete questionnaire responses.
* Total score ≤4 in the pre-test, to preserve data reliability and validity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in knowledge score (mean proportion of correct answers) from baseline to post-intervention. | Baseline and 4 weeks after intervention
  Knowledge assessed using a 16-item questionnaire on the Female Athlete Triad and Relative Energy Deficiency in sport. Each item scored 0-1 and the outcome is a score 0-16 points. A higher scores means better knowledge.

SECONDARY OUTCOMES:
Change in definition questions group | Baseline and 4 weeks after intervention
  Correct answers from the definition questions group. Each question is scored 0-1 and the outcome is a score 0-2 points. A higher scores indicate greater knowledge.
Change in low energy availability questions group | Baseline and 4 weeks after intervention
  Correct answers from the low energy availability questions group. Each question is scored 0-1 and the outcome is a score 0-7 points A higher scores indicate greater knowledge.
Change in menstrual questions group | Baseline and 4 weeks after intervention
  Correct answers from the menstrual questions group. Each question is scored 0-1 and the outcome is a score 0-4 points. A higher scores indicate greater knowledge.
Change in bone health questions group | Baseline and 4 weeks after intervention
  Correct answers from the bone questions group. Each question is scored 0-1 and the outcome is a score 0-3 points. A higher scores indicate greater knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Susana M Gil, MD, PhD, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (1):
- Universidad del Pais Vasco, Leioa, Basque Country, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tam R, Beck KL, Manore MM, Gifford J, Flood VM, O'Connor H. Effectiveness of Education Interventions Designed to Improve Nutrition Knowledge in Athletes: A Systematic Review. Sports Med. 2019 Nov;49(11):1769-1786. doi: 10.1007/s40279-019-01157-y. PMID 31372860
- [Background] Verhoef SJ, Wielink MC, Achterberg EA, Bongers MY, Goossens SMTA. Knowledge on relative energy deficiency in sport among physiotherapists and physicians. Eur J Sport Sci. 2024 Jan 30;24(1):156-63. doi: 10.1002/ejsc.12026. PMCID: PMC11235195.